CLINICAL TRIAL: NCT01487226
Title: A Phase II Trial of Adjuvant Chemotherapy in Patients With Lymph Node Metastasis After Radical Surgery in FIGO Stage IA2-IIA Cervical Cancer
Brief Title: Adjuvant Chemotherapy in Patients With Lymph Node Metastasis After Radical Surgery in Cervical Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korean Gynecologic Oncology Group (Other)
Responsible Party: Principal Investigator, Taek Sang Lee, Principal Investigator, Korean Gynecologic Oncology Group
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KGOG1012
Record Dates: First submitted 2011-12-04; First posted 2011-12-07 (Estimated); Last update posted 2011-12-07 (Estimated); Status verified 2011-12

CONDITIONS: Cervical Cancer
Keywords: Cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Paclitaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: paclitaxel — Paclitaxel 175 mg/m2 over 3 hr Repeat every 3 weeks * 6 cycles
Drug: Cisplatin 50mg/m2 — Cisplatin 50mg/m2
  Repeat every 3 weeks * 6 cycles
  Other Names: Cisplatin

SUMMARY:
Purpose Primary endpoint

* To evaluate the 3-year disease free survival Second endpoints
* To evaluate the 3-year & 5-year overall survival To analyze the toxicity and the quality of life

ELIGIBILITY:
Inclusion Criteria:

* cervical cancer stage Ia2-IIa
* histology; squamous, adeno, adenosquamous subtype
* age; 20∼70 years
* performance status; GOG 0∼2
* no medical illness
* hematologic, renal, hepatic function; normal
* grossly no residual disease
* histologically confirmed lymph nodes metastases
* no parametrial extension and negative resection margin
* number of retrieved lymph nodes; ≥ 20

Exclusion Criteria:

* patients with grade 2 peripheral neuropathy
* patients with uncontrolled infection

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2008-01; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Kaplan-Meier

SECONDARY OUTCOMES:
log-rank test Cox regression analysis

CONTACTS AND LOCATIONS:
Overall Officials: Jong Min Lee, MD, Principal Investigator — Kyung-Hee University East-West Med. Center
Locations (1):
- KGOG, Seoul, South Korea